CLINICAL TRIAL: NCT03205839
Title: Effectiveness of Acceptance-based Self-help for Individuals With Visible Difference and Social Anxiety: a Pilot Randomised Controlled Trial
Brief Title: Acceptance-based Self-help for Individuals With Visible Difference and Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Luke Powell, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151066
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Visible Difference; Acceptance and Commitment Therapy; ACT; Skin Condition; Hair Condition; Craniofacial; Burns
MeSH Terms: conditions — Skin Diseases; Burns

STUDY DESIGN:
Masking Description: Entire study completed online, including randomisation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance-based self-help (Experimental): Participants in this group will receive the self-help booklet.
  Surviving to Thriving: ACT self-help for living well with a visible difference in appearance
  Interventions: Behavioral: Acceptance-based self-help intervention
- Waitlist control group (No Intervention): Participants in this group will be placed onto a waitlist for the four-week intervention period.

INTERVENTIONS:
Behavioral: Acceptance-based self-help intervention — Surviving to Thriving: ACT self-help for living well with a visible difference in appearance.
  A self-help booklet, based upon Acceptance and Commitment Therapy (ACT). The booklet includes some ACT techniques and encourages participants to set themselves behavioural tasks, based upon their values. There is a suggested timetable for participants to navigate through the self-help during the four-week intervention period.
  In addition to the pdf booklet, there are accompanying audio exercises and a lived experience video.
  Other Names: Surviving to Thriving: ACT self-help for living well with...
  Arms: Acceptance-based self-help

SUMMARY:
The acceptance and commitment therapy (ACT) model theoretically fits with treating appearance-related anxiety in individuals with a visible difference. This study examines the effectiveness of an acceptance-based self-help manual for this population.

DETAILED DESCRIPTION:
Individuals with visible difference commonly experience social anxiety due to appearance-related concerns. There are limited resources to help people with appearance-related distress, so internet-provided self-help interventions may be beneficial. A pilot randomised controlled trial will compare the effectiveness of an acceptance-based self-help intervention to a waitlist control group.

We hypothesise (1) the acceptance-based self-help intervention will significantly increase participants' "psychological flexibility", (2) significantly decrease fear of negative evaluation from others and (3) significantly increase their quality of life, compared to the waitlist control group. Data will be collected at two time points only.

General distress (CORE-10) will be collected pre-intervention only to ensure randomisation has been successful. Should the two groups significantly differ in distress, this will be accounted for in subsequent analyses.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who self-identify as having a visible difference to their appearance (such as, but not restricted to: hair and skin conditions, burns, craniofacial conditions, birthmarks, surgical scarring)
* Must self-define as experiencing concerns about social interaction or a loss of social confidence in relation to their visible difference.
* Must be aged 18 years or over
* Must be fluent in English language
* Must have access to a computer and the internet

Exclusion Criteria:

* Currently receiving any form of psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-11-18 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Comprehensive assessment of Acceptance and Commitment Therapy processes | Four weeks
  A general measure of psychological flexibility (and constituent sub-processes) as conceptualized within the ACT model.

SECONDARY OUTCOMES:
Brief Fear of Negative Evaluation Scale II (BFNE-II) | Four weeks
  The BFNE-II is a 12-item revised version of the Brief Fear of Negative Evaluation scale (BFNE; Leary, 1983) used for measuring fears of negative evaluation (e.g., ''I am afraid that others will not approve of me''). Items are rated on a 5-point Likert scale ranging from 0 (not at all characteristic of me) to 4 (extremely characteristic of me). This correlates highly with measures of social anxiety.
Work and Social Adjustment Scale (WSAS) | Four weeks
  Can be used to measure quality of life and functioning impairments in day-to-day life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No current plan, as data this is the first study in the area.